CLINICAL TRIAL: NCT06060834
Title: Impact of a Topical Cosmetic Product Intended to Promote the Health and Beauty of Women's Hair
Brief Title: Impact of a Topical Cosmetic Product on Women's Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of College of Health Sciences, University of Memphis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-FY2024-1
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hair Thinning; Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: pre-post experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Application of product (Experimental): Apply intervention to wet hair on scalp and massage in for 30 seconds after shampooing (if applicable), daily.
  Interventions: Dietary Supplement: Topical Botanical Agent

INTERVENTIONS:
Dietary Supplement: Topical Botanical Agent — Cayenne Pepper, Coconut Water, Kelp, Lemon Juice, Oxynex LM, Potassium Sorbate, Red Palm Oil, Rose Water, Saw Palmetto, vitamin C

SUMMARY:
The proposed pilot study will investigate the impact of a daily topical nutritional product applied to women's hair, specific to perceived hair quality and overall well-being. Hair loss will be measured with a scanning application ("MyHairCounts") , as well as with the 60-second hair comb test. This will be an open-label study with a sample of 15 women and will be used to generate pilot data for future, larger-scale placebo-controlled studies.

DETAILED DESCRIPTION:
Hair loss is commonly experienced by both men and women, with a much greater focus placed on the thinning and loss of hair in women, particularly due to hormonal changes with aging. The loss of hair has biochemical origins and when pronounced, can be a major source of psychological distress which impacts quality of life. Grandview Research Group indicates that the hair and scalp market size is estimated at over $80 billion annually, with hair loss accounting for the majority of share.

Women, in particular, spend significant amounts of money annually on products and treatments specifically focused on hair growth including injections, transplants, and stem cells. While the above treatments are available through a healthcare provider, others are off-the-shelf botanical agents and dietary supplements-some of which have been shown to be effective.

While the anecdotal claims for such products are overwhelmingly positive, very few controlled laboratory studies have been done to investigate the impact of botanical agents on hair beauty and health. While objective outcomes are available (such as the number of hairs lost daily), most individuals focus on the subjective assessments of "beauty" and related items (e.g., shininess of hair, ability to comb and style hair).

The proposed pilot study will investigate the impact of a daily topical nutritional product applied to women's hair, specific to perceived hair quality and overall well-being. Hair loss will be measured with a scanning application ("MyHairCounts") , as well as with the 60-second hair comb test. This will be an open-label study with a sample of 15 women and will be used to generate pilot data for future, larger-scale placebo-controlled studies.

Considering the anecdotal results provided by women who have used the product, coupled with the fact that botanicals and nutritional factors are known to impact hair loss/health, the hypothesis is that women will experience positive results following use, both objectively and subjectively.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 35-70 years
* Subjects should have limp or visibly thin hair, and claim to have experienced mild to moderate hair thinning
* Willing to follow the protocol requirements as evidenced by written informed consent.
* Agree not to use any medication, including vitamins and minerals, or any cosmetic products during or before the course of this study, which are designed to impact hair health.
* Willing to download the MyHairCounts | Hair Loss Prevention | Hair Density Tracking app for use in study assessments.
* Willing to come to the lab for all follow-up visits.
* Have a regular/stable menstrual cycle if not post-menopausal (e.g., 27-32 days).
* Not lactating, pregnant or planning to become pregnant during the study
* Not have any clinically significant medical history (including alopecia), medical finding or an on-going medical or psychiatric condition which in the opinion of the Investigator could jeopardize the safety of the subject, impact validity of the study results or interfere with the completion of study according to the protocol.
* Not have baldness or significant loss of hair, to the extent that the topical product would not remain on the scalp and would run off following application, or if there is such minimal or short hair that an improvement in appearance would not be able to be evaluated.
* Use of any medication or supplement for hair loss, including finasteride, any other 5 α-reductase inhibitor, minoxidil, steroids, or hormonal products, during the 3 months prior to study commencement.
* No history of allergic/sensitivity reactions to product components.
* Must be able to hang loose naturally (unsecured and without hair extensions)

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Hair Density | baseline
  Hair density as determined by "MyHairCounts" application
Hair Density | After 2 weeks of treatment
  Hair density as determined by "MyHairCounts" application
Hair Density | after 1 month of treatment
  Hair density as determined by "MyHairCounts" application
60 second hair count | baseline
  Number of hairs lost when hair is combed for 60 seconds
60 second hair count | After 2 weeks of treatment
  Number of hairs lost when hair is combed for 60 seconds
60 second hair count | after 1 month of treatment
  Number of hairs lost when hair is combed for 60 seconds
Self-assessment of well-being | baseline
  An adaptive visual analog scale will be used to self-assess feelings of confidence, self-consciousness, motivation, and attractiveness/beautifulness on a continuous scale from 0 (not at all) to 10 (extreme).
Self-assessment of well-being | After 2 weeks of treatment
  An adaptive visual analog scale will be used to self-assess feelings of confidence, self-consciousness, motivation, and attractiveness/beautifulness on a continuous scale from 0 (not at all) to 10 (extreme).
Self-assessment of well-being | After 1 month treatment
  An adaptive visual analog scale will be used to self-assess feelings of confidence, self-consciousness, motivation, and attractiveness/beautifulness on a continuous scale from 0 (not at all) to 10 (extreme).
Product assessment | after 1 month of treatment
  An adaptive visual analog scale will be used to self-assess feelings on the smell, ease of use, and self-reported feeling of hair quality using a continuous scale from 1 (not at all) to 10 (Very much).
Self-assessment of hair | baseline
  An adaptive visual analog scale will be used to self-assess feelings on subject's hair (thickness, fullness, shininess, texture, strength, appearance, satisfaction using a continuous scale from 1 (extremely poor) to 10 (Excellent) as well as compliments, split ends on a scale from 1 (Never) to 10 (Very often), ease of styling 1 (very difficult) to 10 (very easy), and speed of hair growth 1 (slow) to 10 (very fast).
Self-assessment of hair | After 2 weeks of treatment
  An adaptive visual analog scale will be used to self-assess feelings on subject's hair (thickness, fullness, shininess, texture, strength, appearance, satisfaction using a continuous scale from 1 (extremely poor) to 10 (Excellent) as well as compliments, split ends on a scale from 1 (Never) to 10 (Very often), ease of styling 1 (very difficult) to 10 (very easy), and speed of hair growth 1 (slow) to 10 (very fast).
Self-assessment of hair | After 1 month of treatment
  An adaptive visual analog scale will be used to self-assess feelings on subject's hair (thickness, fullness, shininess, texture, strength, appearance, satisfaction using a continuous scale from 1 (extremely poor) to 10 (Excellent) as well as compliments, split ends on a scale from 1 (Never) to 10 (Very often), ease of styling 1 (very difficult) to 10 (very easy), and speed of hair growth 1 (slow) to 10 (very fast).

SECONDARY OUTCOMES:
Systolic Blood pressure | baseline
  measured using an automated machine in millimeters of mercury
Diastolic Blood pressure | baseline
  measured using an automated machine in millimeters of mercury
Diastolic Blood pressure | After 2 weeks of treatment
  measured using an automated machine in millimeters of mercury
Systolic Blood pressure | After 2 weeks of treatment
  measured using an automated machine in millimeters of mercury
Diastolic Blood pressure | After 1 month of treatment
  measured using an automated machine in millimeters of mercury
Systolic Blood pressure | After 1 month of treatment
  measured using an automated machine in millimeters of mercury
Heart Rate | baseline
  measured using an automated machine in beats per minute
Heart Rate | After 2 weeks of treatment
  measured using an automated machine in beats per minute
Heart Rate | After 1 month of treatment
  measured using an automated machine in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No